CLINICAL TRIAL: NCT01477606
Title: Phase-II Study Evaluating Midostaurin in Induction, Consolidation and Maintenance Therapy Also After Allogeneic Blood Stem Cell Transplantation in Patients With Newly Diagnosed Acute Myeloid Leukemia Exhibiting a FLT3 Internal Tandem Duplication
Brief Title: Protocol in Acute Myeloid Leukemia With FLT3-ITD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Doehner, Prof. Dr. Hartmut Doehner, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 16-10; 2011-003168-63 (EudraCT Number)
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; FLT3-ITD; midostaurin (PKC412)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Midostaurin (Experimental)
  Interventions: Drug: Midostaurin; Drug: Cytarabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: Midostaurin — Induction therapy: 50 mg, oral, twice daily, starting on day 8, thereafter continuous dosing until 48h before start of subsequent chemotherapy cycle.
  Consolidation therapy: 50 mg, oral twice daily, starting on day 6, thereafter continuous dosing until 48h before start of conditioning therapy for allogeneic HSCT or 48h before start of subsequent consolidation chemotherapy.
  Maintenance therapy:
  50 mg oral twice daily over one year.
  Other Names: PKC412
Drug: Cytarabine — Induction therapy:
  200 mg/m2/day by continuous i.v. infusion on days 1-7 (total dose 1400 mg/m²)
  Consolidation therapy:
  Younger adult patients (18 to 65 yrs): 3 g/m2 by i.v infusion over 3 hours every 12 hours on days 1, 3, and 5 (total dose 18 g/m2).
  Older patients (>65 yrs): 1 g/m2 by i.v. infusion over 3 hours every 12 hours on days 1, 3, and 5 (total dose 6 g/m2).
Drug: Daunorubicin — Induction therapy:
  60 mg/m², by 1-hour i.v. infusion, day 1-3 (total dose 180 mg/m²)

SUMMARY:
This is a phase II, single-arm, open-label, multi-center study in adult patients with Acute Myeloid Leukemia (AML) and FLT3-ITD as defined in inclusion/exclusion criteria.

The primary efficacy object is to evaluate the impact of midostaurin given in combination with intensive induction, consolidation including allogeneic hematopoietic stem cell transplantation and single agent maintenance therapy on event-free survival (EFS) in adult patients with AML exhibiting a FLT3-ITD.

Sample size: 440 patients

The treatment duration of an individual patient is between 18 and 24 months. Duration of the study for an individual patient including treatment (induction, consolidation [chemotherapy or allogeneic SCT], maintenance and follow-up period: Maximum 8 years

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected diagnosis of AML or related precursor neoplasm, or acute leukemia of ambiguous lineage (classified according to the World Health Organization (WHO) 2008 classification)
* Presence of FLT3-ITD assessed in the central AMLSG reference laboratories
* Patients considered eligible for intensive chemotherapy
* WHO performance status of ≤ 2
* Age ≥ 18 years and ≤ 70 years
* No prior chemotherapy for leukemia except hydroxyurea to control hyperleukocytosis (≤ 7 days)
* Non-pregnant and non-nursing. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months)
* Female patients in the reproductive age and male patients must agree to avoid getting pregnant or to father a child while on therapy and for 5 months after the last dose of chemotherapy
* Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control (IUD, tubal ligation, or partner's vasectomy). Hormonal contraception is an inadequate method of birth control
* Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy (while on therapy and for 5 months after the last dose of chemotherapy)
* Signed written informed consent.

Exclusion Criteria:

•AML with the following recurrent genetic abnormalities (according to WHO 2008): AML with t(8;21)(q22;q22); RUNX1-RUNX1T1 AML with inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11 AML with t(15;17)(q22;q12); PML-RARA (or variant translocations with other RARA gene fusions)

* Performance status WHO >2
* Patients with ejection fraction < 50% by MUGA or ECHO scan within 14 days of day 1
* Organ insufficiency (creatinine >1.5x upper normal serum level; bilirubin, AST or ALP >2.5x upper normal serum level, not attributable to AML; heart failure NYHA III/IV; severe obstructive or restrictive ventilation disorder)
* Uncontrolled infection
* Severe neurological or psychiatric disorder interfering with ability of giving an informed consent
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year
* Known positive for HIV; active HBV, HCV, or Hepatitis A infection
* Bleeding disorder independent of leukemia
* No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician and/or other physicians involved in the treatment of the patient about study participation.
* No consent for biobanking.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2012-05; Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Event-free Survival | 8years
  To perform two predefined subgroup analyses in the age-groups 18-60 years and 61-70 years evaluating the impact of midostaurin given in combination with intensive induction, consolidation including allogeneic hematopoietic stem cell transplantation and single agent maintenance therapy on event-free survival (EFS) in adult patients with AML exhibiting a FLT3-ITD.

SECONDARY OUTCOMES:
Rate of complete remission (CR) | Two months
Relapse-free survival | 8 years
overall survival | 8 years
Cumulative incidence of relapse | 8 years
cumulative incidence of death in CR | 8 years
Target (FLT3) inhibition by measuring the FLT3 plasma inhibitory activity | 8 years
  Evaluation of target (FLT3) inhibition by continuous dosing of midostaurin
Quality of life | 5 years
  Quality of life assessed by the EORTC Quality of Life Core Questionnaire (QLQ-C30), supplemented by information on self-assessed concomitant diseases, late treatment effects, and demographics initially, in first CR, after one year,3 and 5 years after initial diagnosis.
Rate of early deaths and hypoplastic deaths (ED/HD) | two months
Death in CR | 8 years
Toxicities | between 18 and 24 months
  Type, frequency, severity (graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 3.0), timing and relatedness of hematological and non-hematological toxicities observed during the different treatment cycles
Impact of allogeneic HSCT | 8 years
  Assessment of the relative impact of allogeneic HSCT analyzed as time-dependent variable on survival endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Doehner, MD, Principal Investigator — University Hospital of Ulm
Locations (55):
- Austria (5):
  - Medizinische Universität Innsbruck, Innsbruck
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - Universitätsklinik für Innere Medizin III Salzburg, Salzburg
  - Hanuschkrankenhaus Wien, Vienna
- Germany (50):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Vivantes Klinikum Neukölln, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - Marienhospital Bochum-Herne, Bochum
  - Medizinische Universitätsklinik Bochum, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Klinikum Darmstadt, Darmstadt
  - Universitätsklinkum Düsseldorf, Düsseldorf
  - Kliniken Essen-Süd, Essen
  - Klinik für Onkologie, Gastroenterologie und Allg. Innere Medizin Esslingen, Esslingen am Neckar
  - Malteser Krankenhaus St. Franziskus Hospital Flensburg, Flensburg
  - Medizinische Universitätsklinik Freiburg, Freiburg im Breisgau
  - MVZ Osthessen, Fulda
  - Klinik der Justus-Liebig-Universität Gießen, Giessen
  - Wilhelm-Anton-Hospital gGmbH Goch, Goch
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - Klinikum Region Hannover GmbH, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - SLK Kliniken Heilbronn GmbH, Heilbronn
  - Universitätskliniken des Saarlandes, Homburg/Saar
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Städtisches Krankenhaus Kiel GmbH, Kiel
  - Caritas Krankenhaus Lebach, Lebach
  - Klinikum Lippe-Lemgo, Lemgo
  - Märkische Kliniken GmbH Lüdenscheid, Lüdenscheid
  - Universitätsklinikum der Otto-von-Guericke Universität Magdeburg, Magdeburg
  - Universitätsklinikum der Johannes Gutenberg-Universität Mainz, Mainz
  - Johannes Wesling Klinikum Minden, Minden
  - Stauferklinikum Mutlangen, Mutlangen
  - Klinikum Schwabing, München
  - Klinikum rechts der Isar der TU München, München
  - Ortenau Klinikum, Offenburg
  - Pius Hospital Oldenburg, Oldenburg
  - Klinikum Oldenburg, Oldenburg
  - Klinikum Passau, Passau
  - Universitätsklinikum Regensburg, Regensburg
  - Caritasklinik St. Theresia Saarbrücken, Saarbrücken
  - Klinikum Stuttgart, Stuttgart
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Klinikum Mutterhaus der Borromäerinnen gGmbH Trier, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Medizinische Universitätsklinik Tübingen, Tübingen
  - University Hospital of Ulm, Ulm
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen, Villingen-Schwenningen
  - Helios Klinikum Wuppertal, Wuppertal

REFERENCES:
- [Derived] Dohner H, Weber D, Krzykalla J, Fiedler W, Wulf G, Salih H, Lubbert M, Kuhn MWM, Schroeder T, Salwender H, Gotze K, Westermann J, Fransecky L, Mayer K, Hertenstein B, Ringhoffer M, Tischler HJ, Machherndl-Spandl S, Schrade A, Paschka P, Gaidzik VI, Theis F, Thol F, Heuser M, Schlenk RF, Bullinger L, Saadati M, Benner A, Larson R, Stone R, Dohner K, Ganser A. Midostaurin plus intensive chemotherapy for younger and older patients with AML and FLT3 internal tandem duplications. Blood Adv. 2022 Sep 27;6(18):5345-5355. doi: 10.1182/bloodadvances.2022007223. PMID 35486475
- [Derived] Schlenk RF, Weber D, Fiedler W, Salih HR, Wulf G, Salwender H, Schroeder T, Kindler T, Lubbert M, Wolf D, Westermann J, Kraemer D, Gotze KS, Horst HA, Krauter J, Girschikofsky M, Ringhoffer M, Sudhoff T, Held G, Derigs HG, Schroers R, Greil R, Griesshammer M, Lange E, Burchardt A, Martens U, Hertenstein B, Marretta L, Heuser M, Thol F, Gaidzik VI, Herr W, Krzykalla J, Benner A, Dohner K, Ganser A, Paschka P, Dohner H; German-Austrian AML Study Group. Midostaurin added to chemotherapy and continued single-agent maintenance therapy in acute myeloid leukemia with FLT3-ITD. Blood. 2019 Feb 21;133(8):840-851. doi: 10.1182/blood-2018-08-869453. Epub 2018 Dec 18. PMID 30563875